CLINICAL TRIAL: NCT05282550
Title: RCT Targeting Cognition in Early Alzheimer's Disease by Improving Sleep With Trazodone (REST)
Brief Title: Targeting Cognition in Early Alzheimer's Disease by Improving Sleep With Trazodone
Acronym: REST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00301426; R01AG071522 (NIH)
Record Dates: First submitted 2022-03-08; First posted 2022-03-16 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: AMCI - Amnestic Mild Cognitive Impairment; Sleep Disturbance
Keywords: AMCI; Slow wave sleep; Trazodone; Cognition
MeSH Terms: conditions — Parasomnias | interventions — Trazodone

STUDY DESIGN:
Intervention Model Description: We will administer trazodone and placebo for 4 weeks each with a 4-week washout.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study drug will be compounded by the Investigational Drug Service (IDS) at Johns Hopkins Bayview Medical Center. The IDS will prepare blind medication using opaque capsules and randomly assign eligible participants to treatment order (ie, starting with trazodone vs. placebo treatment).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trazodone First (Active Comparator): Trazodone (50 mg at bedtime) and then placebo after a 4-week washout period.
  Interventions: Drug: Trazodone; Drug: Placebo
- Placebo First (Placebo Comparator): Placebo and then Trazodone (50 mg at bedtime) after a 4-week washout period.
  Interventions: Drug: Trazodone; Drug: Placebo

INTERVENTIONS:
Drug: Trazodone — 50mg of trazodone administered for 4 weeks.
  Other Names: Desyrel
Drug: Placebo — Placebo administered for 4 weeks.

SUMMARY:
To investigate the effect of trazodone on sleep, hippocampal-dependent memory and hippocampal excitability. The investigators hypothesize that trazodone will improve total sleep time and proportion of time in Slow Wave Sleep (SWS).

DETAILED DESCRIPTION:
The REST trial is a randomized, placebo-controlled, double-blind crossover study of trazodone (50 mg at bedtime) in participants with Amnestic Mild Cognitive impairment (aMCI) and sleep complaints. The investigators will randomize 100 subjects and administer trazodone and placebo for 4 weeks each with a 4-week washout period in between. A 4-week washout period is more than sufficient due to trazodone's elimination half-life of 10-12 hours. The crossover design will facilitate recruitment and enable the use of the subjects as a control without requiring a parallel placebo arm.

ELIGIBILITY:
Inclusion Criteria:

1. Mild Cognitive Impairment (MCI) as defined by Albert et al.2 including subjective memory complaint and/or objective evidence of memory problems;
2. Clinical Dementia Rating (CDR) of 0.5 with a Memory Box score of >=0.5;
3. Evidence of sleep complaints with Pittsburgh Sleep Quality Index score of >5 (a well-validated cutoff observed in >40% of older persons);
4. Memory performance > 1.5 Standard Deviation (SD) below age-and education-matched control subjects on the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) List Recall;
5. Visual and auditory acuity adequate for neuropsychological testing;
6. Good general health with no disease expected to interfere with the study;
7. Able to have Magnetic Resonance Imaging (MRI) scan;
8. Availability of knowledgeable informant (KI)

Exclusion Criteria:

1. Less than 55 years of age to reduce likelihood of including individuals with frontotemporal dementia or non-dementia MCI;
2. Too frail or medically unstable to undergo study procedures;
3. Prior diagnosis of Obstructive Sleep Apnea (OSA) or evidence of moderate-to-severe OSA on baseline Home Sleep Test (HST) as evidenced by an apnea/hypopnea index of >15;
4. Dementia;
5. Cognitive complaints and deficits better explained by other medical/neurologic conditions;
6. Delirium;
7. Allergic to trazodone;
8. Taking sleep medications including trazodone;
9. Current substance abuse;
10. Current major depressive, manic, or acute psychotic episode;
11. Prior diagnosis of significant systemic illness or unstable medical condition which could lead to difficulty complying with the study protocol or represent alternate primary cause of memory problems beyond Alzheimer's Disease (AD) pathology:
12. Lack of available KI;
13. Prior diagnosis of Q wave T wave Corrected for heart rate (QTc) > 470 msec (females) or > 450 msec (males);
14. Inability to provide informed consent

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in total sleep duration between the treatment arms | Baseline and End of study, up to 12 weeks
  Comparison of means of total sleep duration from baseline measured in minutes between trazodone and placebo arm.
Change in Slow Wave Sleep (SWS) duration between the treatment arms | Baseline and End of study, up to 12 weeks
  Comparison of means of SWS from baseline measured in minutes between trazodone and placebo arm.
Change in SWS intensity between the treatment arms | Baseline and End of study, up to 12 weeks
  Comparison of means of SWS intensity measured from baseline in volts squared between trazodone and placebo arm.
Change in sleep onset latency between the treatment arms | Baseline and End of study, up to 12 weeks
  Comparison of means of sleep onset latency from baseline measured in minutes between trazodone and placebo arm.
Change in sleep fragmentation between the treatment arms | Baseline and End of study, up to 12 weeks
  Comparison of means of sleep fragmentation from baseline measured in minutes between trazodone and placebo arm.
Change in self reported sleep measure Pittsburgh Sleep Quality Index (PSQI) between treatment arms | Baseline and End of study, up to 12 weeks
  Comparison of means score for PSQI from baseline between trazodone and placebo arm. A higher score means a worse outcome.
Change in self reported sleep measure Epworth Sleepiness Score (ESS) between treatment arms | Baseline and End of study, up to 12 weeks
  Comparison of means score for ESS from baseline between trazodone and placebo arm. A higher score means a worse outcome.

SECONDARY OUTCOMES:
Change in memory performance between treatment arms | Baseline and End of study, up to 12 weeks
  Comparison of means for memory performance from baseline measured in percent correct between trazodone and placebo arm.
Change in hippocampal activation on Function Magnetic Resonance Imaging (fMRI) measures during memory functioning between treatment arms | Baseline and End of study, up to 12 weeks
  Comparison of means of hippocampal activation on fMRI measures calculated as a beta weight reflecting relative activation during memory functioning from baseline between trazodone and placebo arm. Higher activation suggests a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Barry Greenberg, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The Executive Committee of the study, consisting of the study PIs and the Director of the Data Coordinating Center for this study will oversee the deidentified Individual Participant Data (IPD) sharing. This will include the review of requests for trial data and samples. The Executive Committee will assure that all investigators who receive data and/or specimens are qualified investigators, with research goals consistent with those stated in the consent form. A Material Transfer Agreement (MTA) and/or Data Use Agreement (DUA) will be in place with approved requestors before any transfer of bio-samples or data. Investigators receiving the data and/or samples will be required to cite the grant in any publications generated by the data and to send a copy of all publications to the study team.
Supporting Information: Study Protocol, SAP
Time Frame: 1 year after study completion
Access Criteria: Upon approval of data analytic strategy by study team